CLINICAL TRIAL: NCT06722820
Title: Phase I, First-in-man, Randomised, Placebo-controlled, Single Dose Escalation Study to Investigate the Effects of LPH-5 on Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Parameters in Healthy Participants
Brief Title: Study to Evaluate LPH-5 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lophora (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LPH-5CS01
Record Dates: First submitted 2024-11-19; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Safety Issues; Tolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): LPH-5_dose 1, single dose
  Interventions: Drug: LPH-5; Drug: Placebo
- Cohort 2 (Experimental): LPH-5_dose 2, single dose
  Interventions: Drug: LPH-5; Drug: Placebo
- Cohort 3 (Experimental): LPH-5_dose 3, single dose
  Interventions: Drug: LPH-5; Drug: Placebo
- Cohort 4 (Experimental): LPH-5_dose 4, single dose
  Interventions: Drug: LPH-5; Drug: Placebo
- Cohort 5 (Experimental): LPH-5_dose 5, single dose
  Interventions: Drug: LPH-5; Drug: Placebo
- Cohort 6 (Experimental): LPH-5_dose 6, single dose
  Interventions: Drug: LPH-5; Drug: Placebo

INTERVENTIONS:
Drug: LPH-5 — LPH-5
Drug: Placebo — Placebo

SUMMARY:
This study will explore the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of LPH-5.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, and clinical laboratory evaluations.

Exclusion Criteria:

* Any condition or disease detected during the medical interview/physical examination that could relapse during or immediately after the study, or would render the participant unsuitable for the study, place the participant at undue risk, or interfere with the ability of the participant to complete the clinical study, as determined by the Investigator.
* Have a history of and/or current clinically significant determined by the Investigator
* Consumes cannabis or cannabis-derived compounds more than 3 times per month or has substantial changes in cannabis consumption in the 21 days prior to screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Through study completion, an average of 1 year
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Through study completion, an average of 1 year
Incidence of abnormal clinical laboratory findings in 12-lead ECG parameters, vital signs, and physical examination | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Pharmacokinetics parameters - Cmax | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: maximum plasma concentration (Cmax) (ng/ml)
Pharmacokinetics parameters - tmax | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: time to reach Cmax (tmax) (minutes)
Pharmacokinetics parameters - AUC0-t | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: area under the plasma concentration-time curve (AUC) from zero to the last quantifiable concentration (AUC0-t) (ng/ml x hours)
Pharmacokinetics parameters - AUC0-∞ | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to infinity (AUC0-∞)(ng/ml x hours)
Pharmacokinetics parameters - AUC0-24h | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to 24 hours (AUC0-24h) (ng/ml x hours)
Pharmacokinetics parameters - AUC0-48h | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to 48 hours (AUC0-48h) (ng/ml x hours)
Pharmacokinetics parameters - half life | Time Frame: 0-48 hours
  Plasma PK concentrations including but not limited to: half life (t1/2) (hours)
Pharmacodynamic parameter - assessing the mood and subjective effects of single ascending doses of LPH-5 in healthy participants in questionnaires | Time Frame: 0-48 hours
Pharmacodynamic parameter - Pharmaco-EEG (qEEG) | Time Frame: 0-48 hours
  Power spectral analysis of absolute and/or relative amplitude in the various frequency bands.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Hays, MD, Principal Investigator — Biotrial